CLINICAL TRIAL: NCT00003691
Title: A Randomized Study of Doxorubicin Plus Cisplatin Versus Doxorubicin Plus Cisplatin Plus 3-Hour Paclitaxel With G-CSF Support in Patients With Primary Stage III & IV or Recurrent Endometrial Carcinoma
Brief Title: Combination Chemotherapy With or Without G-CSF in Treating Patients With Stage III, Stage IV, or Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066794; GOG-0177; NCT00698620 (obsolete NCT alias)
Record Dates: First submitted 1999-11-01; First posted 2004-06-24 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2010-09

CONDITIONS: Endometrial Cancer
Keywords: stage III endometrial carcinoma; stage IV endometrial carcinoma; recurrent endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Filgrastim; Cisplatin; Doxorubicin; Paclitaxel

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy consisting of doxorubicin and cisplatin with or without paclitaxel and G-CSF in treating patients who have stage III, stage IV, or recurrent endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the addition of paclitaxel, using filgrastim (G-CSF) support, to standard doxorubicin/cisplatin chemotherapy produces improvement in the frequency of objective response, progression-free survival, or overall survival in patients with stage III, stage IV, or recurrent endometrial carcinoma.
* Compare the toxicities of these two regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive doxorubicin IV over 15-30 minutes, followed immediately by cisplatin IV over 1 hour.
* Arm II: Patients receive doxorubicin and cisplatin as in arm I on day 1. On day 2, patients receive paclitaxel IV over 3 hours. Patients also receive filgrastim (G-CSF) subcutaneously beginning on day 3 and continuing for at least 10 days.

Courses are repeated every 21 days. Treatment continues for up to 7 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 240 patients (120 per arm) will be accrued for this study within 21 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary stage III, stage IV, or recurrent endometrial carcinoma

  * Very poor potential for cure by radiotherapy or surgery alone or in combination
* Measurable disease

  * Disease in an irradiated field as the only site of measurable disease allowed provided there has been clear progression since completion of radiotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* GOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Platelet count at least 100,000/mm^3
* Granulocyte count at least 1,500/mm^3

Hepatic

* SGPT no greater than 3 times upper limit of normal
* Bilirubin normal

Renal

* Creatinine no greater than 1.6 mg/dL

Cardiovascular

* LVEF at least 50% within past 6 months
* No uncontrolled angina
* No third-degree or complete heart block unless a pacemaker is in place

Neurologic

* No serious peripheral neuropathy

Other

* No prior or concurrent malignancy within past 5 years except nonmelanoma skin cancer
* No uncontrolled infection
* No sensitivity to E. coli-derived drug preparations

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior biologic therapy allowed
* No concurrent biologic therapy

Chemotherapy

* No prior cytotoxic chemotherapy, including chemotherapy used for radiation sensitization
* No prior chemotherapy for any prior malignancy

Endocrine therapy

* Prior hormone therapy allowed
* No concurrent hormone therapy

Radiotherapy

* At least 4 weeks since prior radiotherapy to the whole pelvis or to over 50% of the spine

Surgery

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 1998-12; Primary Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gini F. Fleming, MD, Study Chair — University of Chicago
Locations (73):
- United States (72):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Women's Cancer Center, Palo Alto, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Medicine Branch, Bethesda, Maryland
  - Radiation Oncology Branch, Bethesda, Maryland
  - Tufts University School of Medicine, Boston, Massachusetts
  - Memorial Hospital, Worcester, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - Sooner State, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- NCIC-Clinical Trials Group, Kingston, Ontario, Canada

REFERENCES:
- [Background] Farley JH, Tian C, Rose GS, Brown CL, Birrer M, Risinger JI, Thigpen JT, Fleming GF, Gallion HH, Maxwell GL. Chemotherapy intensity and toxicity among black and white women with advanced and recurrent endometrial cancer: a Gynecologic Oncology Group Study. Cancer. 2010 Jan 15;116(2):355-61. doi: 10.1002/cncr.24769. PMID 19924790
- [Background] Moore KN, Tian C, McMeekin DS, Thigpen JT, Randall ME, Gallion HH. Does the progression-free interval after primary chemotherapy predict survival after salvage chemotherapy in advanced and recurrent endometrial cancer?: a Gynecologic Oncology Group ancillary data analysis. Cancer. 2010 Dec 1;116(23):5407-14. doi: 10.1002/cncr.25480. Epub 2010 Aug 24. PMID 20737572
- [Background] McMeekin DS, Filiaci VL, Thigpen JT, Gallion HH, Fleming GF, Rodgers WH; Gynecologic Oncology Group study. The relationship between histology and outcome in advanced and recurrent endometrial cancer patients participating in first-line chemotherapy trials: a Gynecologic Oncology Group study. Gynecol Oncol. 2007 Jul;106(1):16-22. doi: 10.1016/j.ygyno.2007.04.032. PMID 17574073
- [Background] Modesitt SC, Tian C, Kryscio R, Thigpen JT, Randall ME, Gallion HH, Fleming GF; Gynecologic Oncology Group. Impact of body mass index on treatment outcomes in endometrial cancer patients receiving doxorubicin and cisplatin: a Gynecologic Oncology Group study. Gynecol Oncol. 2007 Apr;105(1):59-65. doi: 10.1016/j.ygyno.2006.10.045. Epub 2006 Dec 5. PMID 17150247
- [Background] Maxwell GL, Tian C, Risinger J, Brown CL, Rose GS, Thigpen JT, Fleming GF, Gallion HH, Brewster WR; Gynecologic Oncology Group study. Racial disparity in survival among patients with advanced/recurrent endometrial adenocarcinoma: a Gynecologic Oncology Group study. Cancer. 2006 Nov 1;107(9):2197-205. doi: 10.1002/cncr.22232. PMID 17001661
- [Background] Modesitt S, Tian C, Kryscio R, et al.: Impact of body mass index (BMI) on treatment outcomes in advanced or recurrent endometrial cancer patients receiving doxorubicin/cisplatin chemotherapy: a Gynecologic Oncology Group study. [Abstract] Society of Gynecologic Oncologists, 2006 Annual Meeting on Women's Cancer, March 22-26, 2006, Palm Springs, CA. A-93, 2006.
- [Result] Fleming GF, Brunetto VL, Cella D, Look KY, Reid GC, Munkarah AR, Kline R, Burger RA, Goodman A, Burks RT. Phase III trial of doxorubicin plus cisplatin with or without paclitaxel plus filgrastim in advanced endometrial carcinoma: a Gynecologic Oncology Group Study. J Clin Oncol. 2004 Jun 1;22(11):2159-66. doi: 10.1200/JCO.2004.07.184. PMID 15169803
- [Result] Fleming GF, Brunetto VL, Mundt AJ, et al.: Randomized trial of doxorubicin (DOX) plus cisplatin (CIS) versus DOX plus CIS plus paclitaxel (TAX) in patients with advanced or recurrent endometrial carcinoma: a Gynecologic Oncology Group (GOG) study. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-807, 2002.
- [Result] Huang HQ, Brady MF, Cella D, Fleming G. Validation and reduction of FACT/GOG-Ntx subscale for platinum/paclitaxel-induced neurologic symptoms: a gynecologic oncology group study. Int J Gynecol Cancer. 2007 Mar-Apr;17(2):387-93. doi: 10.1111/j.1525-1438.2007.00794.x. PMID 17362317
- [Result] Grushko TA, Filiaci VL, Mundt AJ, Ridderstrale K, Olopade OI, Fleming GF; Gynecologic Oncology Group. An exploratory analysis of HER-2 amplification and overexpression in advanced endometrial carcinoma: a Gynecologic Oncology Group study. Gynecol Oncol. 2008 Jan;108(1):3-9. doi: 10.1016/j.ygyno.2007.09.007. Epub 2007 Oct 18. PMID 17945336